CLINICAL TRIAL: NCT05170919
Title: An Efficacy Study Comparing Olanzapine and Mirtazapine in the Improvement of Unintentional Weight Loss for Patients with Advanced Stage Cancer
Brief Title: Comparing Olanzapine and Mirtazapine in the Improvement of Unintentional Weight Loss for Patients with Advanced Stage Cancer
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-21-862
Record Dates: First submitted 2021-11-19; First posted 2021-12-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anorexia Nervosa with Significantly Low Body Weight
MeSH Terms: interventions — Mirtazapine; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine (Experimental)
  Interventions: Drug: Olanzapine
- Mirtazapine (Experimental)
  Interventions: Drug: Mirtazapine

INTERVENTIONS:
Drug: Mirtazapine — Patients will be prescribed a dosage of 15 mg per day. Dose will not be escalated.
  Arms: Mirtazapine
Drug: Olanzapine — the participant will be prescribed a dosage of 2.5mg per day if > 65 yrs. and 5 mg/per day if <65 yrs. per day. Per physician discretion, participants are allowed a dose escalation of a maximum of 10mg.
  Arms: Olanzapine

SUMMARY:
To determine whether olanzapine or mirtazapine is more effective in preventing weight loss and appetite loss in cancer patients.

DETAILED DESCRIPTION:
Olanzapine and Mirtazapine have been used in the past few years to attempt to prevent weight and appetite loss in cancer patients. Both have mixed study results and none of the previous studies are of high enough quality to make clinical recommendations. With limited options available, palliative and oncology providers turn to these medications with little evidence. There are no formal studies comparing the two to determine if one is superior to the other, so choices are often made based purely on provider preference. We aim to conduct a study to determine if one of the drugs outperforms the other to guide our standard practice at Englewood Health. This study is being conducted to determine whether olanzapine or mirtazapine is more effective in preventing weight loss and appetite loss in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older

  * Able to provide informed consent
  * Pathologically and/or clinically confirmed diagnosis of advanced cancer
  * At any point of treatment with standard chemotherapy*

    o Scheduled to start, have discontinued or completed, or currently receiving
  * Greater than or equal to 5% unintentional weight loss over the previous 3-6 months, not explained by simple starvation

    o Simple starvation is considered to be excluded when weight loss is not ameliorated by standard nutritional counseling and oral supplementation over a 2-week period).
  * Life expectancy of at least 4 months
  * Able to communicate well and comply with study requirements, including by phone and written logs

    * Patients on Dexamethasone will be allowed

Exclusion Criteria:

* • Abnormal liver function defined as > twice upper limit of normal

  * Elevated QTc

    o EKG performed within 1 year of enrollment will be accepted
  * Total parental nutrition (TPN) or enteral feeds (PEG/PEJ) for >70% of their primary source of daily calorie intake
  * Taking Marinol within 2 week of enrollment onto study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Weight | 6 months
  Patients will have their weight measured every month. A ratio of 5% weight gain or weight stabilization over time will be used to determine if the medication is making an impact.

SECONDARY OUTCOMES:
Quality of Life of patient | 6 months
  Patients will complete a quality of life (QOL) questionnaire provided at each time point. The higher the score, the worse the outcome. Patients will rate their improvement on a scale from 0 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Health, Englewood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No